CLINICAL TRIAL: NCT04315935
Title: Comparison of Analgesic Effect and Prognosis of Butorphanol and Fentanyl in Patients With Mechanical Ventilation: a Prospective, Randomized, Multicenter Clinical Study
Brief Title: Comparison of Analgesic Effect and Prognosis of Butorphanol and Fentanyl in Patients With Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SINGCHN-BUT-IV-1902
Record Dates: First submitted 2020-01-14; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Butorphanol; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- butorphanol group (Experimental): Butorphanol (10-20 μ g / kg / h) analgesia and Propofol (1-4 mg / kg / h) sedation
  Interventions: Drug: Butorphanol and Propofol
- fentanyl group (Active Comparator): Fentanyl (0.7-10 μ g / kg / h) analgesia and Propofol (1-4 mg / kg / h) sedation
  Interventions: Drug: Fentanyl and Propofol

INTERVENTIONS:
Drug: Butorphanol and Propofol — The two groups were given propofol for sedation, BG for butorphanol for analgesia and FG for fentanyl for analgesia
  Arms: butorphanol group
Drug: Fentanyl and Propofol — Fentanyl (0.7-10 μ g / kg / h) analgesia and Propofol (1-4 mg / kg / h) sedation
  Arms: fentanyl group

SUMMARY:
ICU patients often in a strong stress environment. Various invasive procedures such as wound dressing change, sputum suction,Pull out the thoracic duct etc. At the same time, the diseases and environmental factors caused patients anxiety, pain, delirium and even a series of pathophysiological changes which harm life and safety. Fentanyl is an analgesic that acts on central μ receptors, clinical practice had found that fentanyl could exert analgesic effects, while it maybe affect patients' hemodynamics, breathing, and nervous system, which caused hypotension, bradycardia, respiratory depression, delirium and other adverse drug reactions. These reactions prolonged the mechanical ventilation time and duration time of patients in hospital, which impact the treatment effect and prognosis of patients. Butorphanol tartrate is a new type of opioid receptor agonist and antagonist, which can stimulate the κ receptor, and also certain stimulated and antagonised effects on the μ receptor. It can be used for analgesia and sedation in patients of ICU. Previous studies shown that butorphanol can inhibit the inflammatory response and effect myocardial protective. The analgesic effect of butorphanol were equivalent to fentanyl in patients of ICU, and the incidence of nausea and vomiting in participants with butorphanol less than fentanyl. Therefore, the investigators speculate that the analgesia of butorphanol in ICU patients may unexpected effects. However, butorphanol and fentanyl on the analgesic effect and prognosis of patients with mechanical ventilation in ICU are lacking currently, and the investigators no corresponding multi-center clinical study at home and abroad. The research compare to the analgesic effect of butorphanol and fentanyl in critically ill patients with mechanical ventilation. Effects of butorphanol and fentanyl on mechanical ventilation duration, sedation depth, duration time of patients in hospital, complications and mortality in patients with mechanical ventilation. To analyze the high-risk factors affecting the prognosis of patients with mechanical ventilation in ICU. Found more treatment measures for analgesia of patients with mechanical ventilation in ICU.

DETAILED DESCRIPTION:
For enrolled patients, the investigators required that inclusion criteria were informed consent signed.The exclusion criteria were described in detail in the CRF standard. The recruitment of patients into the group were conducted in each sub-center according to Inclusion criteria. After the inclusion of patients will registed relevant information according to the basic data table of patients, disease information table and baseline data table, and then randomly divide the patients into groups by special statistician (CRA/CRO).The relevant data in the clinical study were collected by specialized nurses or data recording team.The daily statistical results need to record and dated by statisticians in order to track the authenticity and reliability of the data. The statistician should communicate with the doctor in charge about the situation out the trial plan during the study. If there is any change in the test plan, it is necessary to mark the measures and reasons for the change in detail, and sign the signature and date of the statistician and the responsible doctor in the statistical table of the day. The recorded data of the study should be updated with electronic documents. Statistical recorder of data need to make weekly summary, summarize and submit the statistical data of last month at each sub-research center at the beginning of each month, then the lead hospital will summarize and analyze the data.As for the problems beyond the experimental schemes in the research process, each branch center needs to discuss with the lead center. Every three months, progress meetings will be held to discuss various problems in clinical research and to unify standards for related problems to ensure the smooth progress of clinical research and the true reliability of experimental results. SAS 9.4 software was used for statistical analysis. The analysis content included subject distribution description, baseline index balance analysis, efficacy analysis and safety analysis.The significance level of the statistical test was α=0.05. In the safety analysis, the incidence of adverse events and adverse reactions was calculated and the specific conditions of all subjects with adverse events were listed. The list of vital signs and normal abnormalities in laboratory examination before and after medication was described, and the specific conditions of subjects with abnormal conditions before and after treatment and abnormal conditions before and after treatment were listed in detail.After completing the statistical analysis, the statistical analyst should record the data and submit it to the main researcher of the experiment to fill with the general analysis report. All cases, whether observation or shedding, should be completed in accordance with the requirements of "case report form". The case report form were copied three copies with without carbon copy. After the completion of data entry, the sponsor (the first copy), the unit in charge of the clinical research (the second copy) and the clinical research unit (the third copy) shall file it respectively.

ELIGIBILITY:
Inclusion Criteria:

1. aged >= 18 years, 18kg / m2 < BMI < 30 kg / m2;
2. patients with invasive mechanical ventilation (refer to the clinical application guide of mechanical ventilation [2006];
3. the expected ventilation time was >= 24h, and the ventilation time was < 48h;
4. sign the informed consent voluntarily and participate in the research. -

Exclusion Criteria:

1. known allergy to any study drug;
2. for chronic pain of grade 3 or above in the World Health Organization, strong opioids, such as morphine, are often used. Recently, opioids are used for analgesia through spinal cord catheter, epidural or any other regional block;
3. the American Society of anesthesiologists (ASA) classified the fifth grade patients (on the verge of death);
4. nerve injury or brain organic pathological changes;
5. participate in clinical research in the past 30 days;
6. pregnancy or lactation;
7. the researcher thinks it is not suitable to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic score, | Maintain target analgesia score (CPOT<3) from 100% time to 80% time
  Analgesia score (CPOT < 3 points)
sedative score | Maintain target analgesia score (CPOT<3) from 100% time to 80% time
  APACHE II score, SOFA score,
Total dosage of butorphanol， fentanyl，propofol; | Maintain target analgesia score (CPOT<3) from 100% time to 80% time
  The specific dosage of butorphanol, fentanyl and propofol,

SECONDARY OUTCOMES:
Major indicators affecting the prognosis of patients in ICU | From day 1 to day 30
  pulling time, ICU stay time, invasive mechanical ventilation time, length of stay, 30 day mortality

OTHER OUTCOMES:
Incidence of adverse reactions | From day 1 to day 30
  The percentages of delirium, respiratory depression, hypotension, tachycardia, pneumonia, intestinal obstruction, renal failure, wound infection, and nausea/vomiting were recorded in different groups,

CONTACTS AND LOCATIONS:
Overall Officials: Quansheng Q Du, doctor, Principal Investigator — Hebei People's Hospital
Locations (1):
- Hebei People's Hospital, Hebei, Hebei, China

IPD SHARING:
Plan to Share IPD: No
The clinical study data of this project were owned by the participating research center. For other researchers who need data, the results of the study can be understood through the literature published later.